CLINICAL TRIAL: NCT06362798
Title: Effect of Support for Low-Income Mothers of Preterm Infants on Parental Caregiving in the Neonatal Intensive Care Unit (NICU)
Brief Title: Effect of Support for Low-Income Mothers of Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Margaret Parker, Professor of Pediatrics, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Study00001150; 1R01HD109293-01 (NIH); 6-23FY-0012 (Other Grant/Funding Number: March of Dimes)
Record Dates: First submitted 2024-03-22; First posted 2024-04-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth; Low; Birthweight, Extremely (999 Grams or Less)
MeSH Terms: conditions — Premature Birth; Birth Weight

STUDY DESIGN:
Intervention Model Description: Two-arm single-blind 1:1 randomized controlled trial of financial transfers ($160 per week) versus usual care. Mothers in the intervention arm will access videos that explain the impact of the cash on their availability for benefits and social supports. They will also be able to ask questions to a benefits counselor about how the transfers affect their benefits during the trial.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Enrolled mothers who are assigned to the intervention group will be informed to not discuss the financial transfers with anyone on the NICU care team (i.e., physicians, nurses, etc.)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Transfers (Experimental): Mothers assigned to the intervention group will be informed that they are eligible to receive financial transfers $160/week on a "CuddleCard" debit-card with a one- time "label" or scripted message that states: "This money is intended to help you to spend more time visiting and caring for your infant(s) in the NICU." Financial transfers will begin 1 week after birth or when the mother is discharged (whichever comes later) until the infant is discharged, except in cases where the hospitalization lasts beyond 42 weeks corrected age.
  Interventions: Other: Financial Transfers
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Financial Transfers — Mothers assigned to the intervention group will be informed that they are eligible to receive financial transfers $160/week on a debit-card with a one-time "label" or scripted message that states: "This money is intended to help you to spend more time visiting and caring for your infant(s) in the NICU." Financial transfers will begin 1 week after birth or when the mother is discharged (whichever comes later) until the infant is discharged, except in cases where the hospitalization lasts beyond 42 weeks corrected age.
  Arms: Financial Transfers

SUMMARY:
Preterm birth is a leading cause of childhood mortality and developmental disabilities. Socioeconomic disparities in the incidence of preterm birth and morbidities, mortality, and quality of care for preterm infants persist. An important predictor of the long-term consequences of preterm birth is maternal presence during the prolonged infant hospitalization (weeks to months) in the neonatal intensive care unit (NICU). Mothers who visit the NICU can pump breast milk, directly breastfeed and engage in skin-to-skin care, which facilitates breast milk production and promotes infant physiologic stability and neurodevelopment. Low-income mothers face significant barriers to frequent NICU visits, including financial burdens and the psychological impact of financial stress, which hinder their participation in caregiving activities. The investigators will conduct an randomized controlled trial (RCT) to test the effectiveness of financial transfers among 420 Medicaid - eligible mothers with infants 24 - 34 weeks' gestation in four level 3 NICUs: Boston Medical Center (BMC) in Boston, Massachusetts, UMass Memorial Medical Center (UMass) in Worcester, Massachusetts, Baystate Medical Center in Springfield, Massachusetts, and Grady Memorial Hospital in Atlanta, Georgia. Mothers in the intervention arm will receive usual care enhanced with weekly financial transfers and will be informed that these transfers are meant to help them spend more time with their infant in the NICU vs. a control arm (usual care). We received supplemental funding to extend analyses to include extended postpartum maternal health outcomes. The original sample size of 420 remains the basis for the parent trial's primary and secondary NICU caregiving outcomes, while the supplemental funding (effective January 2026) enables analysis of secondary maternal health outcomes up to 12 months postpartum using an expanded analytic cohort. The primary hypothesis is that financial transfers can enable economically disadvantaged mothers to visit the NICU, reduce the negative psychological impacts of financial distress, and increase maternal caregiving behaviors associated with positive preterm infant health and development.

ELIGIBILITY:
Inclusion Criteria:

* Mother is eligible for Medicaid insurance.
* Has an infant or infants born 24 0/7-34 1/7 weeks gestation.
* Mother's baby is cared for at one of the four enrolling study sites located in Massachusetts or Georgia.
* Mother is eligible to breastfeed (per hospital criteria).

Exclusion Criteria:

* Mother is not English- or Spanish-speaking.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Provision of breast milk (proportion) | From NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Proportion of nursing shift-total enteral intake that is maternal breast milk fed via gavage tube or bottle.
Provision of skin-to-skin care | From NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Proportion of nursing shifts where mother performs skin-to-skin care for at least one hour.

SECONDARY OUTCOMES:
Duration of mother's milk expression | From NICU admission through to 12 months postpartum
  Months of milk expression via direct breastfeeding or pumping.
Gestational weight-for-age | Extracted from medical records 1-2 weeks after discharge from the NICU
  Change in sex-specific gestational weight-for-age z-score while admitted to the NICU.
Gestational length-for-age z-score | Extracted from medical records 1-2 weeks after discharge from the NICU
  Change in sex-specific gestational length-for-age z-score while admitted to the NICU.
Gestational head circumference | Extracted from medical records 1-2 weeks after discharge from the NICU
  Change in sex-specific gestational head circumference z-score while admitted to the NICU.
Necrotizing enterocolitis (NEC) | Extracted from medical records 1-2 weeks after discharge from the NICU
  Experienced NEC during NICU stay according to Vermont Oxford Network (VON) definition; criteria: yes/no.
Late-onset bacterial or fungal sepsis (LOS) | Extracted from medical records 1-2 weeks after discharge from the NICU
  Experienced with LOS during NICU stay according to Vermont Oxford Network (VON) definition; criteria: yes/no.
NICU Visitation | From NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Proportion of nursing shifts where mother is present in the NICU.
Postpartum Bonding | Measured in the post-discharge survey within 4-8 week of infant discharge
  Score of mother-infant bonding assessed inspired by the Postpartum Bonding Questionnaire, where participants rate their agreement of statements on Likert scales ranging from 0 (always) to 5 (never); scores range from 0 to 50, with higher scores indicating more bonding challenges.
Provision of breast milk (volume) | From NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Milliliters of nursing shift-total enteral intake that is maternal breast milk fed via gavage tube or bottle.
Breastfeeding episode | From NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Occurrence of direct breastfeeding episode during each nursing shift.
Maternal physical health | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of self-reported Short Form Health Survey -1 Physical Health Item; assesses participants' perception of their current physical health. Lower score indicates worse perceived physical health.
Maternal mental health (anxiety) | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of self-reported 10-item Perceived Stress Scale (PSS-10); assesses the perceived stress levels experienced in terms of overstrain, unmanageability, and unpredictability in the past month. Higher score indicates worse outcome.
Maternal mental health (depression) | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of the Edinburgh Postnatal Depression Scale (EPDS), a 10-item self-report measure of postpartum depression (ranges from 0-30) with a higher score indicating worse depressive symptoms. The EPDS was developed to assist health professionals in detecting mothers suffering from postpartum depression (PPD).
Reaction Time Attention Network Test-Revised (ANT-R). | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Average response time across all trials to assess overall speed of responses. Lower scores indicate faster reaction times and better attentional performance.
Accuracy Performance Attention Network Test-Revised (ANT-R). | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Proportion of accurate responses on the ANT-R. Higher scores indicate higher accurate responses.
Reaction Time Psychomotor Vigilance Task | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Average reaction time across trials, assessing overall speed and vigilance. Lower scores indicate quicker reaction times and heightened vigilance.
Accuracy Psychomotor Vigilance Task | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks)
  Percentage of correct responses out of the total number of trials on the Psychomotor Vigilance Task (PVT). Higher scores indicate higher accurate responses.
Happiness | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score on Happiness Indicator from Integrated Values Surveys; assesses the overall and current perceived level of happiness experienced; with a 4-point scale from 0 (Not at all happy) to 3 (Very Happy). Higher score indicates better perceived level of happiness.
Life satisfaction | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of the Life Satisfaction Scale Item; assesses participants' perception of their current overall life satisfaction; with a 4-point scale from 0 (Very Satisfied) to 3 (Not At All Satisfied), and was reverse-coded such that higher scores indicate better perceived life satisfaction.
Sleep | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of Sleep Quality Score (SQS) with 7-Day Recall; evaluates the overall quality of sleep. Core components include sleep duration, ease of falling asleep, frequency of waking during the night (excluding bathroom visits), early waking, and sleep refreshment. The respondent marks an integer score from 0 to 10, according to the following five categories: 0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent. Higher score indicates better perceived sleep quality.
Routine postpartum care | Measured at post-discharge (4-8 weeks after infant discharge from NICU); 6 months postpartum; 12 months postpartum
  Number of routine postpartum follow-up visits attended by mom.
Financial distress | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of financial stress during the NICU stay based on two metrics: difficulty in paying bills and remaining money at the end of the week. Scoring for each question is summed to create an overall financial distress score, ranging from 0 to 8. Higher score indicates higher financial distress.
Financial hardship | Measured within one week of discharge form the NICU; post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of financial hardships experienced during the NICU stay, including using up all savings, taking out loans, borrowing from friends, incurring debt, being threatened by eviction, or having a shut-off of an energy utility. Scoring for each question is yes/no and is summed to create an overall score that ranges between 0 and 6.
Food insecurity | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score of Food Insecurity Screening Tool; assesses the risk of food insecurity (availability and affordability) in households based on questions derived from the U.S. Household Food Security Survey Module. Response options include: "Often True," "Sometimes True," "Never True". An affirmative response on either item will be considered to be positive for food insecurity.
Housing instability | Measured within one week of discharge form the NICU; post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Number of moves family has made since their child's birth.
Housing insecurity | Measured within one week of discharge form the NICU; post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score on housing insecurity scale; assesses participants' worry that they may not have stable housing in the next 2 months. Likert scales ranging from 0 (not at all worried) to 3 (very worried). Higher scores indicate greater levels of housing insecurity.
Transportation insecurity | Measured biweekly from NICU admission to discharge or 42 weeks corrected gestational age, whichever comes earlier (maximum of 18 weeks); post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Score on transportation insecurity item; assesses participants' experience of transportation-related issues affecting their ability to visit the NICU. Likert scales ranging from 0 (never) to 3 (always). Higher scores indicate greater levels of transportation insecurity.
Length of stay | Measured within one week of discharge form the NICU
  The total number of days from infant admission to discharge from the hospital.
Mother readmission between 4-8 weeks post-discharge | Measured between 4-8 weeks after discharge of infant from NICU
  Any mother readmission to the hospital after her initial discharge.
Baby readmission between 4-8 weeks post-discharge | Measured between 4-8 weeks after discharge of infant from NICU
  Any infant readmission to the hospital after initial discharge.
Mother emergency department visit post-discharge | Measured at post-discharge survey (4-8 weeks after infant discharge from NICU); 6 months postpartum; 12 months postpartum
  The number of emergency department visits by the mother in the postpartum period.
Baby emergency department visit weeks post-discharge | Measured at post-discharge survey (4-8 weeks after infant discharge from NICU); 6 months postpartum; 12 months postpartum
  The number of emergency department visits by the infant after discharge.
Sleep position | Measured between 4-8 weeks after discharge of infant from NICU
  Mothers report of exclusive infant supine position to sleep in the last two weeks.
Sleep location | Measured between 4-8 weeks after discharge of infant from NICU
  Mothers report exclusively using the room-sharing sleep method, where the infant sleeps in the same room as an adult but on a separate crib or sleep surface, without bed-sharing, in the last two weeks.
Breastfeeding expression continuation | Measured between 4-8 weeks after discharge of infant from NICU
  Mothers report of breastfeeding continuation.
Skin-to-skin care knowledge | Measured within one week of discharge form the NICU
  Mothers report of knowledge about Skin-to-skin (STS) care based on 4 questions. Scored as a count variable that ranges between 0 and 4.
Breastfeeding knowledge | Measured within one week of discharge form the NICU
  Mothers report of knowledge about breastfeeding based on 7 questions. Scored as a count variable that ranges between 0 and 7.
Perception of hospital experience | Measured between 4-8 weeks after discharge of infant from NICU
  Assesses mothers' overall perception of hospital experience and hospital services during their stay, using a scale from 0 (worst hospital possible) to 10 (best hospital possible).
Life's Essential 8 (LE8) behavioral cardiovascular health score | Measured at pre-discharge; post-discharge (4-8 weeks, where all components are available); 6 months postpartum; 12 months postpartum
  Composite score (0-100) based on four behavioral components: diet quality, physical activity, sleep health, and nicotine exposure, scored according to American Heart Association Life's Essential 8 criteria.
Primary care utilization in the postpartum period | Measured at post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Number of visits with a primary care provider for routine or sick care.
Adherence to recommended care for chronic conditions | Measured at post-discharge (4-8 weeks); 6 months postpartum; 12 months postpartum
  Self-reported adherence to recommended postpartum care for chronic conditions (hypertension, diabetes, and mental health), including medication adherence and engagement with healthcare providers for condition management.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Parker, MD, Principal Investigator — UMass Memorial Health; Margaret McConnell, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (4):
- United States (4):
  - Children's Healthcare of Atlanta and Emory University, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts

REFERENCES:
- [Derived] McConnell M, Alsager A, Fuchu P, Sriprasad S, Simoncini L, Drainoni ML, Cordova-Ramos EG, Pena MM, Madore L, Kalluri NS, Silverstein M, Schofield H, Farah MJ, Fink G, Parker MG. CuddleCard: Protocol for a randomized controlled trial evaluating the effect of providing financial support to low-income mothers of preterm infants on parental caregiving in the neonatal intensive care unit (NICU). BMC Pediatr. 2025 May 15;25(1):383. doi: 10.1186/s12887-025-05621-9. PMID 40375176